CLINICAL TRIAL: NCT02983877
Title: Improving Medication Adherence in Hypertensive Individuals With Bipolar Disorder
Brief Title: Medication Adherence in Hypertensive Individuals With Bipolar Disorder
Acronym: iTAB-CV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Jennifer Levin, Associate Professor, Case Western Reserve University
Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: HL132364
Record Dates: First submitted 2016-11-29; First posted 2016-12-06 (Estimated); Results first posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Hypertension; Bipolar Disorder
MeSH Terms: conditions — Hypertension; Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Following a 30 day run-in period, Stage 1 of the iTAB-CV intervention will be introduced. A member of the study team will conduct an interview in order to customize iTAB-CV for each participant at the baseline session. In the first month of iTAB-CV, participants will receive alternating daily texts with psychoeducational and motivational content once daily and a daily mood rating request to both monitor their mood and to determine engagement with the iTAB-CV intervention. In the second stage of iTAB-CV, participants will receive daily texts which will include medication reminders, contextual cues, and immediate reinforcement for medication taking behavior in addition to the content from stage 1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iTAB-CV (Experimental): In the Individualized Texting for Adherence Building-CV (iTAB-CV) Stage 1, participants will receive alternating daily texts with educational and motivational content on treatment for high blood pressure and bipolar disorder, and a daily mood rating request to both monitor their mood and to determine adherence to iTAB-CV intervention. Stage 1 will last one month.
  In the Individualized Texting for Adherence Building-CV (iTAB-CV) Stage 2, participants will receive daily texts which will include medication reminders, contextual cues, and immediate reinforcement for medication taking behavior in addition to the content from Stage 1. Stage 2 will last one month.
  Interventions: Behavioral: iTAB-CV

INTERVENTIONS:
Behavioral: iTAB-CV — Stage 1 of the intervention will be introduced. Researchers will conduct an interview in order to customize iTAB-CV for each participant at the baseline session. In the first month, participants will receive alternating daily texts with educational and motivational content and a daily mood rating request to both monitor their mood and to determine adherence to the intervention.
  In the second stage for the following month, participants will receive daily texts which will include medication reminders, contextual cues, and immediate reinforcement for medication taking behavior in addition to the content from stage 1.
  Other Names: Individualized Texting for Adherence Building-CV

SUMMARY:
This study will test an adherence intervention (iTAB-CV) delivered via interactive text messaging which first targets behavioral intent and then adds cues/reminders and reinforcement to form the habit of taking antihypertensives in non-adherent individuals with BD. Thirty eight individuals with BD and HTN being treated with evidence-based antihypertensive agents and mood stabilizing or antipsychotic medications who are non-adherent with their HTN medicine will be enrolled.

This study uses a prospective cohort design with participants serving as their own control. Investigators will test the iTAB-CV intervention quantitatively for feasibility and acceptability as well as for efficacy in increasing adherence to antihypertensives, decreasing systolic blood pressure, and increasing adherence to BD medication.

DETAILED DESCRIPTION:
This study will test an adherence intervention (iTAB-CV) delivered via interactive text messaging which first targets behavioral intent and then adds cues/reminders and reinforcement to form the habit of taking antihypertensives in non-adherent individuals with BD. Thirty eight individuals with BD and HTN being treated with evidence-based antihypertensive agents and mood stabilizing or antipsychotic medications who are non-adherent with their HTN medicine will be enrolled.

This study uses a prospective cohort design with participants serving as their own control. Investigators will test the iTAB-CV intervention quantitatively for feasibility and acceptability as well as for efficacy in increasing adherence to antihypertensives, decreasing systolic blood pressure, and increasing adherence to BD medication.

All study participants will be followed for a 3-month period. iTAB-CV, delivered via mobile phone, is intended to be a brief adjunct to standard primary care and mental health treatment. All individuals will continue to receive treatment as usual with their regular provider(s). Individuals who meet eligibility criteria will have a 30 day run-in period in which their medication adherence will be measured with TRQ and MEMS but without an additional intervention. Following the run-in period, Stage 1 of the iTAB-CV intervention will be introduced. Researchers will conduct an interview in order to customize iTAB-CV for each participant at the baseline session. In the first month of iTAB-CV, participants will receive alternating daily texts with psychoeducational and motivational content once daily and a daily mood rating request to both monitor their mood and to determine engagement with the iTAB-CV intervention. In the second stage of iTAB-CV, participants will receive daily texts which will include medication reminders, contextual cues, and immediate reinforcement for medication taking behavior in addition to the content from stage 1.

Assessments that include evaluation of treatment adherence, psychiatric symptoms, self-efficacy for medication taking behavior, illness beliefs, medication attitudes, and habit strength for both antihypertensive and BD medications will be conducted at four time points over a 3-month time period (screening, baseline/week 4, week 8, and week 12). Blood pressure will be measured at each of the four contacts. Individuals who drop out of the intervention, and who agree, will be followed up with outcomes assessments over the same 3-month time period that they would have been evaluated had they remained in the study.

About one month after study completion, a member of the research team will call each participant and ask questions about their bipolar and blood pressure medication taking habits.

ELIGIBILITY:
Inclusion criteria:

1. Participants will have a clinical diagnosis of BD for at least 2 years as determined by a standardized diagnostic interview, the Mini-International Neuropsychiatric Interview (MINI) (52)
2. Have stage 1 or 2 HTN with a systolic pressure ≥130
3. Carry a diagnosis of HTN per patient self-report ≥ 6 months prior to enrollment
4. Have been prescribed at least one regularly scheduled antihypertensive medication for ≥ 3 months since diagnosis
5. Have self-reported poor adherence to antihypertensive medication defined as at least 20% of days with missed doses for at least one antihypertensive in either the past week or past month as identified by the Tablets Routine Questionnaire (TRQ).
6. Be able to participate in psychiatric interviews

Exclusion criteria:

1. Unable or unwilling to participate in psychiatric interviews. This will include individuals, who may be too psychotic to participate in interviews/rating scales
2. Unable or unwilling to give written, informed consent to study participation
3. Under the age of 21
4. In the interest of patient safety, individuals who are at high immediate risk for suicide will be excluded from study participation. The suicide risk assessment will be informed by standardized assessments of psychiatric symptoms and the Mini-International Neuropsychiatric Interview (MINI). In the event that a potential study participant is determined to be at high risk for suicide, that individual will not be enrolled and the study staff will immediately implement procedures for the safety of the individual. Once such individuals are deemed stable, they may be once again considered for inclusion in the research.
5. Individuals who are monolingual, non-English speaking will be excluded. Given the relatively small sample size in the proposed study, it would not be practical to conduct sub-group analyses. Also, the study assessment tools and the texting intervention are not available in other languages and would be impractical to develop. Based upon our BD adherence work, which drew upon a population similar to the proposed trial, there were no potential subjects who were excluded from the studies due to inability to speak English.
6. Illiterate participants will be excluded because reading is an essential skill required to complete self-report questionnaires administered during the study as well as to respond to the text messages which make up the intervention.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Levin, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center and Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levin JB, Sajatovic M, Rahman M, Aebi ME, Tatsuoka C, Depp C, Cushman C, Johnston E, Cassidy KA, Blixen C, Eskew L, Klein PJ, Fuentes-Casiano E, Moore DJ. Outcomes of Psychoeducation and a Text Messaging Adherence Intervention Among Individuals With Hypertension and Bipolar Disorder. Psychiatr Serv. 2019 Jul 1;70(7):608-612. doi: 10.1176/appi.ps.201800482. Epub 2019 Apr 17. PMID 30991908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty eight individuals with bipolar disorder (BD) and hypertension (HTN) being treated with evidence-based antihypertensive agents and mood stabilizing or antipsychotic medications who are nonadherent with their HTN medicine will be enrolled by referral. This phase uses a prospective cohort design with participants serving as their own control.
Pre-assignment Details: After providing informed consent, all participants will undergo screening followed by a 30-day run-in period in which adherence will be measured using eCAP and self-report. During the 30-day run-in period, participants will continue to receive care as usual and serve as their own control with no intervention.
Groups:
- iTAB-CV: In the Individualized Texting for Adherence Building-CV (iTAB-CV) Stage 1, participants will receive alternating daily texts with educational and motivational content on treatment for high blood pressure and bipolar disorder, and a daily mood rating request to both monitor their mood and to determine adherence to iTAB-CV intervention. Stage 1 lasts one month.
  Stage two of iTAB-CV includes the addition of customized context cues/reminders and immediate reinforcement for medication taking behavior in addition to 1 daily motivational mood rating. The number of texts per day will be determined based on the number of times a day that medications are prescribed (up to four a day). Stage two lasts one month.
Period: Overall Study
Arm/Group | iTAB-CV
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- iTAB-CV: In the Individualized Texting for Adherence Building-CV (iTAB-CV) Stage 1, participants will receive alternating daily texts with educational and motivational content on treatment for high blood pressure and bipolar disorder, and a daily mood rating request to both monitor their mood and to determine adherence to iTAB-CV intervention.
  iTAB-CV Stage 1: Stage 1 of the intervention will be introduced. Researchers will conduct an interview in order to customize iTAB-CV for each participant at the baseline session. In the first month, participants will receive alternating daily texts with educational and motivational content and a daily mood rating request to both monitor their mood and to determine adherence to the intervention.
Arm/Group | iTAB-CV
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.53 (9.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 28
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 38
Years of education [Mean (Standard Deviation); unit: years] | 13.18 (2.69)
Employment [Count of Participants; unit: Participants]
  Full time/homemaker | 1
  Part time | 3
  Unemployed, but expected to work by self or others | 6
  Disabled | 28
Bipolar disorder type [Count of Participants; unit: Participants] — Baseline diagnostic assessment of type of bipolar disorder. Bipolar I Disorder is defined by manic episodes that last at least 7 days, or by manic symptoms that are so severe that the person needs immediate hospital care. Usually, depressive episodes occur as well, typically lasting at least 2 weeks. Episodes of depression with mixed features (having depression and manic symptoms at the same time) are also possible.
  Bipolar II Disorder is defined by a pattern of depressive episodes and hypomanic episodes, but not the full-blown manic episodes described above.
  Participants
    Bipolar Disorder Type I | 28
    Bipolar Disorder Type II | 10
Age of hypertension diagnosis [Mean (Standard Deviation); unit: years] | 36.95 (15.66)
Age of bipolar disorder diagnosis [Mean (Standard Deviation); unit: years] | 31.95 (13.46)
hypertension-related hospitalizations [Median (Full Range); unit: occurrences] — Number of hypertension-related hospitalizations over participant's lifetime. Population: Nineteen people endorsed having at least one hypertension-related hospitalization in their lifetime. Therefore, the median number of how many hospitalizations they had are based solely on those 19, to eliminate skewing of results of everyone who answered 0 lifetime hypertension-related hospitalizations.
  occurrences
    number analyzed (Participants) | 19
    (all) | 3.16 [1 to 15]
substance use-related hospitalizations [Median (Full Range); unit: occurrences] — Number of hospitalizations related to substance use over the participant's lifetime. Population: Twelve people endorsed having at least one hypertension-related hospitalization in their lifetime. Therefore, the median number of how many hospitalizations they had are based solely on those 12, to eliminate skewing of results of everyone who answered 0 lifetime substance use-related hospitalizations.
  occurrences
    number analyzed (Participants) | 12
    (all) | 3.00 [1 to 10]
History of physical abuse [Count of Participants; unit: Participants]
  Yes | 20
  No | 18
History of sexual abuse [Count of Participants; unit: Participants]
  Yes | 20
  No | 18
Mental illness in the family [Count of Participants; unit: Participants]
  Yes | 30
  No | 8
Smokes cigarettes [Count of Participants; unit: Participants]
  Yes | 23
  No | 15
Median number of cigarettes smoked per day [Median (Full Range); unit: cigarettes per day] — Population: Twenty-three people endorsed being a cigarette smoker. Therefore, the median number of how many cigarettes smoked per day is based solely on those 23, to eliminate skewing of results of everyone who answered they are not cigarette smokers.
  cigarettes per day
    number analyzed (Participants) | 23
    (all) | 6.00 [1 to 20]
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.15 (9.40)

OUTCOME MEASURES:

1. Primary Outcome: Change in Adherence to Anithypertensives Based on Tablets Routine Questionnaire (TRQ)
Description: This self-report measure identifies non-adherence for the past 7 days (Scott & Pope, 2002a, 2002b), by measuring the percentage of days with missed doses of a given medication. Adherence will be assessed for each regularly scheduled antihypertensive that has been prescribed for ≥ 3 months. For individuals who are on more than one medication, an average TRQ will be calculated for all antihypertensive medications. PRN medications will not be included.
Time Frame: change from Screen (Week 0) to V2 (week 12)
Population: Baseline descriptives
Measure: Mean (Standard Deviation); unit: percentage of days with missed doses
Groups:
- Whole Sample: These analyses were run on the entire sample as a whole, N= 38.
Arm/Group | Whole Sample
Number analyzed (Participants) | 38
percentage of days with missed doses
  Screen visit antihypertensive TRQ (past week) | 42.86 (23.15)
  V2 (week 12) antihypertensive TRQ (past week) | 21.24 (17.95)
Statistical Analysis 1: Comparison: Whole Sample; Test type: Superiority; p < 0.001, Friedman test; 3 degrees of freedom

2. Secondary Outcome: Change in Systolic Blood Pressure
Time Frame: change from Screen (Week 0) to V2 (week 12)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Whole Sample
Number analyzed (Participants) | 38
mmHg
  Screen visit systolic blood pressure | 144.81 (15.46)
  V2 (12 week) systolic blood pressure | 136.02 (17.77)
Statistical Analysis 1: Comparison: Whole Sample; Test type: Superiority; p < 0.001, ANOVA; 3 degrees of freedom

3. Secondary Outcome: Change in Adherence to Bipolar Medication Based on the Tablets Routine Questionnaire (TRQ)
Description: This self-report measure identifies non-adherence for the past 7 days (Scott & Pope, 2002a, 2002b), by measuring the percentage of days with missed doses of a given medication. Adherence was assessed for each evidence-based BD regularly scheduled maintenance medication (lithium, anticonvulsant, antipsychotic) prescribed for ≥ 3 months. For individuals who were on more than one medication, an average TRQ was calculated for all BD medications. According to our study team's recent work, the correlation between a single "index" drug and all BD drugs was 0.95 providing support for measuring one medication as proxy for medication adherence (M. Sajatovic et al., 2015). PRN medications were not included.
Time Frame: change from Screen (Week 0) to V2 (week 12)
Population: Missing data for one participants (i.e. n= 37).
Measure: Mean (Standard Deviation); unit: percentage of days with missed doses
Groups:
- Whole Sample: These analyses were run on the entire sample as a whole. For this measure, two participants were missing data so the total N=36 instead of 38.
Arm/Group | Whole Sample
Number analyzed (Participants) | 37
percentage of days with missed doses
  Screen visit bipolar medication TRQ (past week) | 43.95 (27.27)
  V2 (12 week) bipolar medication TRQ (past week) | 25.86 (23.01)
Statistical Analysis 1: Comparison: Whole Sample; Test type: Superiority; p < 0.001, Friedman test; 3 degrees of freedom

4. Secondary Outcome: Change in Adherence to Antihypertensives Based on the Electronic Monitoring Device (eCAP)
Description: Study participants will be given an eCAP device for one of their pill bottles, which will record time/date of bottle opening. eCAP will be used for the antihypertensive medication that the patient missed the most frequently in the past week (in the case of multiple antihypertensive medications missed the same proportion of times, the medication dosed most often will be chosen). A dose will be counted as "taken" if the bottle is opened within six hours of the prescribed time. We will calculate a percent of doses taken by dividing the number of times the bottle is opened by the number of times it should have been opened as per the prescription.
Time Frame: change from Baseline (Week 4) to V2 (week 12)
Measure: Mean (Standard Deviation); unit: percentage of medications missed
Arm/Group | Whole Sample
Number analyzed (Participants) | 38
percentage of medications missed
  Baseline visit antihypertensive eCAP (past week) | 37.70 (28.19)
  V2 (12 week) antihypertensive eCAP (past week) | 34.75 (28.88)
Statistical Analysis 1: Comparison: Whole Sample; Test type: Superiority; p = 0.89, ANOVA; 2 degrees of freedom

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- iTAB-CV: Participants received alternating daily texts with educational and motivational content on treatment for high blood pressure and bipolar disorder, and a daily mood rating request to both monitor their mood and to determine adherence to iTAB-CV intervention.
Arm/Group | iTAB-CV
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 9/38
Other Adverse Events (participants affected / at risk) | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iTAB-CV (N=38)
stomach pain (Gastrointestinal disorders) | 1 (3)
Voluntary alcohol rehab at VA (Social circumstances) | 1 (1)
diverticulitis (Gastrointestinal disorders) | 1 (1)
kidney stones (Renal and urinary disorders) | 1 (2)
suicidal thoughts (Psychiatric disorders) | 2 (2)
high blood pressure (Blood and lymphatic system disorders) | 1 (1)
hyperglycemia (Blood and lymphatic system disorders) | 1 (1)
swollen legs (General disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT02983877/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT02983877/ICF_001.pdf